CLINICAL TRIAL: NCT04532437
Title: Computer-based Skin Aging Simulation for Skin Cancer Prevention: A Pilot Study
Brief Title: Computer-based Skin Aging Simulation for Skin Cancer Prevention
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2020-00963; sp20Maul3
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Skin Aging
Keywords: skin cancer prevention; skin aging simulation; UV-exposure; skin analysis photo system; VISIA® photo analysis system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: artificial intelligence-based skin aging simulation — Photographs of the volunteers' facial skin will be taken in the Department of Dermatology at baseline using a modern skin analysis photo system (VISIA®, Canfield Scientific, Parsippany, NJ, USA) and afterwards a simulation of the participants' facial skin aging will be performed with the VISIA® photo analysis System.
Other: electronic questionnaire 1 — Electronic questionnaire about current sun-related knowledge and protective behaviours via link with smartphone before and after the skin aging simulation.
Other: electronic questionnaire 2 — Participants report their perception of the interventions and their motivation for improved sun protection by completing an electronic questionnaire after the skin aging simulation.

SUMMARY:
This pilot study is to assess the knowledge, attitudes, and practices regarding skin cancer prevention in young adults and to determine the impact of artificial intelligence-based simulation of facial skin aging on their attitudes regarding skin cancer prevention.

DETAILED DESCRIPTION:
In young adulthood an increasing UV-exposure often starts because of the belief that tanning increases attractiveness]. Raising awareness and educating students and adults regarding practices for skin cancer prevention are critical since skin cancer is increasing rapidly worldwide. Skin cancer preventive interventions for adolescents are needed to improve their motivation for sun safety behavior. This pilot study is to assess the knowledge, attitudes, and practices regarding skin cancer prevention in young adults and to determine the impact of artificial intelligence-based simulation of facial skin aging on their attitudes regarding skin cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* healthy female volunteers
* written,Institutional Review Board (IRB)/ Independent Ethics Committee (IEC)-approved informed consent.

Exclusion Criteria:

* skin diseases requiring medical therapy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy female volunteers aged 18-35 years, e.g. medical students of the University Basel, who do not have any skin diseases requiring medical therapy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale (VAS) score regarding importance of UV- protection | before and after the skin aging simulation (each scoring session will take about 15-20 minutes)
  Change in VAS score regarding importance of UV- protection (0 = not important; 10 = extremly important)
Change in VAS score regarding rating of personal exposure to UV radiation | before and after the skin aging simulation (each scoring session will take about 15-20 minutes)
  Change in VAS score regarding rating of personal exposure to UV radiation (0 = no exposure; 10 = very high exposure)

SECONDARY OUTCOMES:
Questionnaire asking for reduction of UV- exposure (yes/no) | after the skin aging simulation (each scoring session will take about 15-20 minutes)
  Questionnaire asking for reduction of UV- exposure (yes/no)
Questionnaire asking for intensification of UV protection measures (yes/ no) | after the skin aging simulation (each scoring session will take about 15-20 minutes)
  Questionnaire asking for intensification of UV protection measures (yes/ no)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Valeska Maul, Dr. med., Principal Investigator — Department of Dermatology, University Hospital Basel
Locations (1):
- Department of Dermatology, University Hospital Basel, Basel, Switzerland